CLINICAL TRIAL: NCT02740790
Title: Immunogenicity and Safety of Recombinant Human Papillomavirus Bivalent(Type 16 and 18) Vaccine (Yeast) in Healthy Females
Brief Title: Immunogenicity and Safety of Human Papillomavirus (HPV)-16/18 Vaccine in Healthy Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 311-HPV-1002
Record Dates: First submitted 2016-02-18; First posted 2016-04-15 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Human Papillomavirus
Keywords: Human papillomavirus; vaccine; cervical infection; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- HPV vaccine 1 (Experimental): 300 women between 9-17 yeas of age, receiving 0,2,6 month-schedule experimental HPV vaccines
  Interventions: Biological: HPV vaccine
- Placebo 1 (Placebo Comparator): 300 women between 9-17 yeas of age, receiving 0,2,6 month-schedule Placebo.
  Interventions: Biological: Placebo
- HPV vaccine 2 (Experimental): 120 women between 18-26 yeas of age, receiving 0,2,6 month-schedule experimental HPV vaccines
  Interventions: Biological: HPV vaccine
- HPV vaccine 3 (Experimental): 180 women between 27-45 yeas of age, receiving 0,2,6 month-schedule experimental HPV vaccines
  Interventions: Biological: HPV vaccine
- Placebo 2 (Placebo Comparator): 120 women between 18-26 yeas of age, receiving 0,2,6 month-schedule Placebo.
  Interventions: Biological: Placebo
- Placebo 3 (Placebo Comparator): 180 women between 27-45 yeas of age, receiving 0,2,6 month-schedule Placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPV vaccine — Subjects were planned to receive HPV vaccine 0.5ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule
  Arms: HPV vaccine 1; HPV vaccine 2; HPV vaccine 3
Biological: Placebo — Subjects were planned to receive three doses of the placebo control 0.5ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule
  Arms: Placebo 1; Placebo 2; Placebo 3

SUMMARY:
Evaluate immunogenicity and safety of recombinant human papillomavirus bivalent ( types 16 and 18 ) vaccine ( Yeast )in different age group. And evaluate persistence of immune response in 9-17years age group. To demonstrate that 9-17years age group was non-inferior to 18-26 years age group and 27-45 years age group in terms of immunogenicity.

DETAILED DESCRIPTION:
This study is a multi-centre, randomized, blinded, placebo controlled study. The study vaccine is recombinant human papillomavirus bivalent (types 16 and 18) vaccine (Yeast), the placebo is aluminium phosphate diluent.

After informed and received the consent of participants/guardians, 1200 healthy females aged 9-45 will be enrolled into three age groups: 9-17, 8-26, 27-45. With the proportion of 1:1, vaccine group and placebo group will receive injection of 0.5ml of vaccine or placebo diluent.

Participants will be injected of vaccine or placebo on a three-dose schedule (0, 2, 6 months). After each inoculation, the immediate reaction will be observed for 30 minutes, and the local and systemic reaction will be systematically observed for 7 days. After the first inoculation, adverse event will be collected until one month after the final inoculation, while serious adverse event will be collected until 6 months after the final inoculation. For every participants, blood samples will be collected before the first inoculation (month 0), one month after the final inoculation (month 7), 6 months after the final inoculation (month 12) to detect the neutralizing antibody of HPV type 16 and 18, and proceed safety and immunogenicity analysis. For participants in 9-14 age group who received the vaccine, neutralizing antibody will also be detected in month 24, 36 and 48 to examine the immune persistency. Meanwhile, some participants will be chosen to study the deviation of gene expression after the vaccination and the association of that with the neutralizing antibody level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female between, and including, 9 and 45 years of age at the time of the first vaccination
* Provide legal identification for for the sake of recruitment
* Be able to understand and sign informed consent prior to enrollment (For subjects below the legal age of consent, informed consent must be signed by parent(s)/legal guardian(s) in addition).
* Subject must be not pregnant at the enrollment and agree to using adequate contraceptive precautions within 7 months.

Exclusion Criteria:

* History of cervical cancer
* Previous administration of any HPV vaccine
* History of severe allergic reaction requiring medical intervention (such as oral and throat swelling, difficulty breathing, hypotension or shock)
* History of allergic to vaccine, or to any ingredient of vaccine.
* History of epilepsy, seizures or convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose.
* History of asthma, thyroidectomy, angioneurotic edema, diabetes or malignant
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* Acute disease or chronic disease acute exacerbation 7 days prior to vaccination
* Administration of immunoglobulins and/or any blood products within 3 months, or administration of any live attenuated vaccine within 28 days, or administration of any subunit or inactivated vaccines within 14 days.
* Fever or axillary temperature> 37.0 °C before vaccination
* During menstrual period, breastfeeding, pregnancy(pregnancy test positive), or planned pregnant within 7 month
* History of hypertension, physical examination systolic blood pressure> 150mmHg and/or diastolic blood pressure> 100mmHg
* Abnormal laboratory tests parameters
* Any clinical significant disease or findings during study screening that, in the opinion of the Investigator may interfere with the study

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The neutralizing antibody responses of HPV 16/18 after vaccination by measuring Geometric Mean Titer (GMT). | 1 month after vaccination

SECONDARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of any solicited local or systemic reactions | 7 days after each vaccine dose
Occurrence, intensity and relationship to vaccination of any solicited local or systemic reactions | 6 months after finish vaccinations
The durability of neutralizing antibody responses of HPV 16/18 after vaccination. | 48 months after finish vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Rong-cheng Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No